CLINICAL TRIAL: NCT02444091
Title: Cyclophosphamide in Myalgic Encephalopathy/ Chronic Fatigue Syndrome (ME/CFS). Part A: an Open Label Phase-II Study With Six Intravenous Cyclophosphamide Infusions Four Weeks Apart, and Follow-up for 12 Months
Brief Title: Cyclophosphamide in Myalgic Encephalopathy/ Chronic Fatigue Syndrome (ME/CFS)
Acronym: CycloME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Kavli Foundation (Unknown); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTS-7-2015; 2014-004029-41 (EudraCT Number)
Record Dates: First submitted 2015-03-25; First posted 2015-05-14 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2019-12

CONDITIONS: Chronic Fatigue Syndrome (CFS); Myalgic Encephalomyelitis (ME)
Keywords: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis (ME); Cyclophosphamide; Immunomodulatory treatment; CFS
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide (Experimental): Cyclophosphamide, intravenous infusions four weeks apart. Six infusions in total. First infusion: 600 mg/m2. Infusions 2 to 6: 700 mg/m2
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide intravenous infusions four weeks apart, in total six infusions. First infusion: cyclophosphamide 600mg/m2. Infusions 2 to 6: cyclophosphamide 700 mg/m2 . Follow-up for 12 months.

SUMMARY:
Significant clinical improvements of ME/CFS symptoms were observed in two patients with long-standing ME/CFS who received adjuvant chemotherapy including cyclophosphamide for breast cancer, also in one ME/CFS patient who received chemotherapy including iphosphamide for Hodgkin lymphoma.

Three pilot ME/CFS patients were thereafter treated with six intravenous infusions four weeks apart, in two of these with a significant clinical response.

The hypothesis is that a subset of ME/CFS patients have an activated immune system, and that ME/CFS symptoms may be alleviated by treatment with cyclophosphamide as intravenous pulse infusions four weeks apart, six infusions in total.

The purpose of the present study is to treat ME/CFS patients with cyclophosphamide as intravenous pulse infusions four weeks apart, six infusions in total. The effects on ME/CFS symptoms and tolerability/side effects during 12 months follow-up will be registered, and additional tests will be performed to objectively register changes in physical ability during follow-up. Studies to investigate possible large vessel endothelial dysfunction and skin microvascular dysfunction will be performed before start of intervention and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ME/CFS according to "Canadian" criteria (2003)
* Duration of ME/CFS at least 2 years
* Mild/Moderate, Moderate, Moderate/Severe and Severe ME/CFS may be included
* Age 18-65 years
* Signed informed consent

Exclusion Criteria:

* Patients with fatigue who do not comply by the diagnostic "Canadian" criteria (2003) for ME/CFS
* Duration of ME/CFS less than 2 years
* Mild ME/CFS
* Very severe ME/CFS (bedridden requiring help for all tasks)
* Patients where the workup uncovers other pathology as possible cause of symptoms
* Pregnancy or breast feeding
* Previous malignant disease (except basal cell carcinoma of skin and cervical carcinoma in situ/dysplasia)
* Previous long-term systemic treatment with immunosuppressive agents (e.g. azathioprine, ciclosporin, mycophenolate mofetil). Except steroid treatment for e.g. obstructive lung disease or autoimmune diseases such as e.g. ulcerative colitis
* Serious endogenous depression
* Lack of ability to complete the study including follow-up
* Reduced renal function (creatinine > 1.5 x UNL)
* Reduced liver function (bilirubin or transaminases > 1.5 x UNL)
* Known hypersensitivity to cyclophosphamide or metabolites
* Reduced bone marrow function
* Ongoing cystitis or urinary tract obstruction
* Known HIV positivity, previous hepatitis B or hepatitis C, or reason to suspect other ongoing and clinically relevant infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Fatigue score, selfreported | Within 12 months follow-up
  Selfreported Fatigue score is registered every second week, always compared to baseline, as the mean of the four symptoms: "Post-exertional malaise", "Fatigue", "Need for rest", Daily functioning" (scale 0-6, in which 3 is unchanged from baseline). Mean Fatigue scores for the time intervals 0-3, 3-6, 6-9 and 9-12 months are recorded for each patient. Changes in selfreported Fatigue scores from baseline to the mean values in each of the time intervals 0-3, 3-6, 6-9 and 9-12 months follow up, will constitute the primary endpoint.
  Responses for the primary endpoint will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Overall response | Within 12 months follow-up
  Overall response is recorded as the effect on ME/CFS symptoms during 12 months follow-up. The overall response is not predefined to a specific time interval during follow-up, but is defined as mean Fatigue score at least 4.5 for at least 6 consecutive weeks for moderate response, and mean Fatigue score at least 5.0 for at least 6 consecutive weeks for major response. Single response periods and the sum of response periods during 12 months follow-up will be recorded.
  Overall response will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.

SECONDARY OUTCOMES:
Short Form-36 (SF-36) | Recorded at baseline, and at 3, 6, 9 and 12 months follow-up.
  SF-36 (ver 1.2) is completed by patients at baseline, and at 3, 6, 9, 12 months follow-up. Changes in Physical health summary score, Physical function, and "Mean of five subdimensions" (Physical function, Bodily pain, Vitality, Social function, General health) from baseline to each of the time points 3, 6, 9 and 12 months follow-up are recorded and constitute secondary endpoints. Secondary endpoints will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Physical activity (Sensewear armband) | Recorded at baseline, at 7-9 months, and at 11-12 months
  The patients' physical activity level, in a home setting for 7 consecutive days, is recorded using Sensewear armbands, with registration at baseline and repeated in the time interval 7-9 months follow-up, and in the interval 11-12 months. Changes from baseline to analysis during the time intervals 7-9 months and 11-12 months, for mean number of steps per 24h, maximum number of steps per 24h, mean duration per 24h with activity level at least 3.5 METs, max duration per 24h with activity level at least 3.5 METs, are recorded. Changes in Physical activity will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Cardiopulmonary exercise tests for two following days | At baseline, and repeated at 7-9 months, and 11-12 months
  For patients who can tolerate exercise, cardiopulmonary exercise tests will be performed for two consecutive days, at baseline, and repeated in the time intervals 7-9 months, and 11-12 months. A programmed ramp-protocol is used. Oxygen-uptake and work load (Watt) day 2, at maximum effort and at anaerobic threshold, will be recorded and used for comparison to oxygen-uptake and work load with repeated tests after 7-9 and 11-12 months. Changes from baseline to repeated exercise tests after 7-9 and 11-12 months will be analyzed.
Self-recorded Function level | At baseline, and at 3, 6, 9 and 12 months follow-up
  Self-recorded "Function level" (scale 0-100, compared to healthy state, according to a set of examples) are registered every second week. Mean "Function level" for the time intervals 0-3, 3-6, 6-9, 9-12 months are calculated. The changes in selfreported "Function level", from baseline to the mean value during each of the the time intervals 0-3, 3-6, 6-9, 9-12 months constitute secondary endpoints.
  Changes in Self-reported Function level will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Fatigue Severity Scale | Baseline, 3, 6, 9 and 12 months
  Fatigue Severity Scale (FSS) is completed by patients at baseline and at 3, 6, 9, 12 months. The changes in FSS from baseline to 3, 6, 9 and 12 months constitute secondary endpoints.
  Changes in Fatigue severity scale will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Longest continuous response duration | Within 12 months follow-up
  The longest duration of continuous self-reported Fatigue score ≥ 4,5 (for at least 6 consecutive weeks) within 12 months follow-up.
  The longest response duration will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response and for the group with previous rituximab intervention with clinical response but later relapse, and also for all 40 included patients together.
Sustained clinical response at 12 months | Assessment at end of follow-up (12 months)
  The fraction of patients with sustained clinical response (defined as Fatigue score of at least 4.5) at 12 months, constitute a secondary endpoint.
  Sustained clinical response at 12 months will be recorded separately for the group of (at least) 25 ME/CFS patients not given rituximab previously, for the group with previous rituximab intervention for ME/CFS with no clinical response, and for the group with previous rituximab intervention with clinical response but later relapse, and for all included patients together.
Safety and tolerability | Continuously within the study period of 12 months
  Safety will be assessed by interim history, physical examination, and laboratory assessments every four weeks the first six months, thereafter at 6, 9 and 12 months follow-up. Adverse events will be graded according to the Common Toxicity Criteria for Adverse Effects (NCI-CTCAE, version 4.0). Number of patients with any grade, or severe (≥ grade 3 NCI-CTCAE version 4.0) toxicity will be reported, as a measure of tolerability and safety.
  Adverse Events may include include hair loss, vomiting, diarrhea, jaundice, leukopenia, anemia, thrombocytopenia, infections, allergic reactions and hemorrhagic cystitis, disturbed ovarian function. The investigators will also collect information on possible toxicity after the formal 12 months study period.

CONTACTS AND LOCATIONS:
Overall Officials: Mella Olav, MD, PhD, Principal Investigator — Haukeland University Hospital; Øystein Fluge, MD, PhD, Study Director — Haukeland University Hospital
Locations (1):
- Dept. of Oncology, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Fluge O, Bruland O, Risa K, Storstein A, Kristoffersen EK, Sapkota D, Naess H, Dahl O, Nyland H, Mella O. Benefit from B-lymphocyte depletion using the anti-CD20 antibody rituximab in chronic fatigue syndrome. A double-blind and placebo-controlled study. PLoS One. 2011;6(10):e26358. doi: 10.1371/journal.pone.0026358. Epub 2011 Oct 19. PMID 22039471
- [Background] Fluge O, Mella O. Clinical impact of B-cell depletion with the anti-CD20 antibody rituximab in chronic fatigue syndrome: a preliminary case series. BMC Neurol. 2009 Jul 1;9:28. doi: 10.1186/1471-2377-9-28. PMID 19566965
- [Derived] Rekeland IG, Fossa A, Lande A, Ktoridou-Valen I, Sorland K, Holsen M, Tronstad KJ, Risa K, Alme K, Viken MK, Lie BA, Dahl O, Mella O, Fluge O. Intravenous Cyclophosphamide in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. An Open-Label Phase II Study. Front Med (Lausanne). 2020 Apr 29;7:162. doi: 10.3389/fmed.2020.00162. eCollection 2020. PMID 32411717